CLINICAL TRIAL: NCT05880433
Title: The Effects of Mydriatic Eye Drops on Cerebral Blood Flow and Oxygenation in Retinopathy of Prematurity Examinations: A Prospective Observational Trial
Brief Title: The Effects of Mydriatic Eye Drops in Retinopathy of Prematurity Examinations
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Didem Arman, Associate Professor, Istanbul Training and Research Hospital
Other Study IDs: IstanbulTRH-DArman-001
Record Dates: First submitted 2023-05-09; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Retinopathy of Prematurity; Mydriasis; Neonatal Disease; Analgesic Adverse Reaction
Keywords: Cerebral blood flow; Cerebral oxygenation; Mydriatic eye drops; Doppler ultrasonography; Retinopathy of prematurity; NIRS; Neonate
MeSH Terms: conditions — Retinopathy of Prematurity; Mydriasis; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before Eye drop instillation: For pupil dilatation, one drop of 2.5% phenylephrine hydrochloride and 0.5% tropicamide was instilled three times at 5 minute intervals, 1 hour before the exam. All infants were fed 1 hour before instillation of drops and infants were swaddled before the procedure.
  Interventions: Device: NIRS(INVOS 5100; Covidien Somanetics, Troy, MI
- After Eye drop instillation: The same participiants investigated after eye drop instillation
  Interventions: Device: NIRS(INVOS 5100; Covidien Somanetics, Troy, MI

INTERVENTIONS:
Device: NIRS(INVOS 5100; Covidien Somanetics, Troy, MI — NIRS (Near Infrared Spectroscopy) is a non-invasive, bedside device that measures the concentration of oxygenated and deoxygenated hemoglobin in tissue, providing information about tissue oxygenation. Its working mechanism is based on the ability of light with wavelengths between 700-1000 nm to penetrate up to 8 cm into the skin and brain tissue. It offers continuous information about tissue oxygenation in different regions using probes attached to the skin. While pulse oximeters indicate arterial oxygen saturation, they are insufficient in detecting tissue-level hypoxia. Therefore, NIRS, being a painless method, is frequently used in the monitoring of newborns in the intensive care unit.

SUMMARY:
Retinopathy of prematurity (ROP) is a retinal disorder of preterm neonates and a potential cause of blindness. As early diagnosis and treatment preserve vision, very low birth weight infants must be screened for ROP. Mydriatic eye drop administration is essential to perform funduscopic evaluations. The most commonly used mydriatic drops for pupil dilatation are 0.5-1.0% tropicamide and/or 0.5-1.0% phenylephrine or 0.2-1.0% cyclopentolate. Phenylephrine, an alpha-1 sympathomimetic agonist, is readily absorbed from conjunctival mucosa and has a potent systemic vasopressor effect. Tropicamide causes cycloplegia by inhibition of ciliary muscle contraction and has a short acting para-sympatholytic effect.

Systemic absorption of mydriatic eye drops has been associated with cardiovascular, respiratory and gastrointestinal adverse effects. Systemic side effects include apnea, desaturation, increased heart rate and blood pressure, delayed gastric emptying, and feeding intolerance. The data about the effects of mydriatics on cerebral blood flow and tissue oxygenation are sparse. Cerebral blood flow autoregulation depends in part on the adrenergic and cholinergic control of cerebral vasculature, but whether mydriatics have an effect on cerebral haemodynamics is unknown. Near-infrared spectroscopy and Doppler ultrasonography (US) are non-invasive methods commonly used for neuromonitorization in NICUs. The regional blood flow changes measured using Doppler US have been reported to be associated with cerebral oxygenation and indicate a high correlation with NIRS in newborns.

The aim of this study was to evaluate the effects of mydriatic eye drops on cerebral oxygenation and blood flow in preterm infants by NIRS and Doppler US.

ELIGIBILITY:
Inclusion Criteria:

* Babies born at gestational age less than 34 weeks and/or birth weight below 2000 grams.

Infants undergoing their first retinopathy examination.

Exclusion Criteria:

* Congenital anomaly

  * Continued mechanical ventilation support
  * Having pain from a different cause and/or requiring concurrent analgesic use
  * Sedation analgesia administered within the last 24 hours
  * Hemodynamically unstable
  * Intraventricular hemorrhage, neurological dysfunction
  * Receiving anticonvulsant therapy.

Ages: 28 Days to 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sixty two infants with a gestational age below 34 weeks and/or with a birth weight of less than 2000 g. were included in the study. The infants who underwent the initial retinopathy screening exam and did not need any respiratory support at the time of the examination were included. The neonates with congenital anomaly, sepsis, hemodynamic instability and intraventricular hemorrhage were excluded.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
NIRS | Data were started to get recorded 60 minutes before the instillation of eye drops for pupil dilation. The recording was continued uninterruptedly till 1 hour after the instillation through study completion, an average of 2 hours.
  Absolute change in rScO2 after mydriatic eye drops instillation with NIRS
Doppler US measurements | The initial and second assessment were conducted before the application and at the 60th minute of instillation of the first drop, respectively - an average of 2 hours.
  Absolute change in MCA blood flow after mydriatic eye drops instillation with Doppler USG

SECONDARY OUTCOMES:
Changes in heart rate (beats per minute) | starting 60 minutes before and after mydriatic eye drop instillation,through study completion, an average of 2 hours.
  Heart rate was recorded continuously, starting 60 minutes before and after mydriatic eye drop instillation.
Changes in blood pressure | Starting 60 minutes before and after mydriatic eye drop instillation,through study completion, an average of 2 hours.
  Mean arterial pressure values was recorded for every 5 minutes, starting 60 minutes before and after mydriatic eye drop instillation,through study completion, an average of 2 hours.
Changes in oxygen saturation. | Starting 60 minutes before and after mydriatic eye drop instillation,through study completion, an average of 2 hours.
  Oxygen saturation was recorded continuously, starting 60 minutes before and after mydriatic eye drop instillation, through study completion, an average of 2 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- IstanbulTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No